CLINICAL TRIAL: NCT00402142
Title: Phase II Study of Autologous Myeloid Dendritic Cells as a "Cellular Adjuvant" for a Therapeutic HIV-1 Vaccine in Early Stage HIV-1+ Patients (DCV-2).
Brief Title: Dendritic Cell Vaccine in HIV-1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Felipe Garcia, Principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCV-02/MANON07
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
Keywords: HIV Infection; Dendritic cell vaccine; Autologous virus; Heat inactivated; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pulsed dendritic cells untreated patients (Active Comparator): Untreated patients receiving a dendritic cell based vaccine pulsed with autologous heat iactivated virus
  Interventions: Biological: Dendritic cell vaccine
- non pulsed dendritic cells untreated patients (Placebo Comparator)
  Interventions: Biological: non pulsed dendritic cell untreated patients
- pulsed dendritic cell treated patient (Active Comparator): treated patients will be immunized with a dendritic cell vaccine pulsed with heat inactivated autologous virus immediately before art interruption
  Interventions: Biological: pulsed dendritic cell vaccine
- pulsed dendritic cell in treated patients (Active Comparator): patients will be immunized with a dendritic cell vaccine pulsed with heat inactivted autologous virus immediately after interruption of art
  Interventions: Biological: dendritic cell vaccine
- non pulsed dendritic cells (Placebo Comparator)
  Interventions: Biological: non pulsed dendritic cell vaccine

INTERVENTIONS:
Biological: Dendritic cell vaccine — 107 DC subcutaneous 3 doses every 2 weeks
  Arms: Pulsed dendritic cells untreated patients
Biological: non pulsed dendritic cell untreated patients — 107 DC subcutaneous 3 doses every 2 weeks
  Arms: non pulsed dendritic cells untreated patients
Biological: pulsed dendritic cell vaccine — 107 DC subcutaneous 3 doses every 2 weeks
  Arms: pulsed dendritic cell treated patient
Biological: dendritic cell vaccine — 107 DC subcutaneous 3 doses every 2 weeks
  Arms: pulsed dendritic cell in treated patients
Biological: non pulsed dendritic cell vaccine — 107 DC subcutaneous 3 doses every 2 weeks
  Arms: non pulsed dendritic cells

SUMMARY:
1. To study the efficacy of a therapeutic HIV vaccine consisting of autologous myeloid dendritic cells pulsed ex vivo with high doses of inactivated autologous HIV-1, in HIV-1 infected patients in a very early stages of the disease (CD4 > 450 x 10 6 /L).
2. To analyze the HIV-1 humoral and cellular immune responses induced by this immune-based therapy.

DETAILED DESCRIPTION:
Our group has reported recently the first human trial of 4 therapeutic immunizations at six-week intervals with autologous monocyte-derived dendritic cells (MD-DC) loaded with heat-inactivated autologous HIV in 12 HIV infected patients who had been receiving highly active antiretroviral therapy (HAART) since early chronic infection. Autologous HIV was concentrated from plasma (1,500 ml) obtained by plasmapheresis after a 3-month HAART interruption (STOP1) performed 78 weeks before therapeutic immunizations, and HAART was discontinued again (STOP2) after therapeutic immunization. There was a decrease of set-point plasma viral load (PVL) >= 0.5 log after 24 weeks off HAART in 4 out of 12 patients. In addition, we observed a significant lengthening in mean doubling time of PVL rebound (p= 0.01), and significant decreases in the area under the curve of PVL rebound (p= 0.02) and in the mean peak PVL (p= 0.004) during the 12 weeks after STOP 2 compared with STOP1. This virological response was associated with a weak but significant increase in HIV-1 specific CD4 lymphoproliferative response, and with changes in HIV-1 specific CD8+ T-cell responses in peripheral blood and in lymphoid CTL cells after immunization. In lymphoid tissue, we also observed a trend towards a better control of HIV-1 replication coupled with an increase of CD4+ and CTL cells. No significant virological or immunological changes occurred in controls. We show that a therapeutic vaccine with autologous MD-DC pulsed with heat inactivated autologous HIV-1 is feasible, safe and well tolerated and elicited weak and transient cellular immune responses against HIV, associated with a partial and transient control of HIV replication in some patients.

we hypothesized that a DC vaccine pulsed with higher amount of autologous virus obtained by culture could be more effective than the vaccine we used.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* CD4 > 450 x 10 6 /L
* baseline VL >10,000 c/ml before any HAART
* Part I, patients off HAART at least during 6 months
* Part II, Patients on HAART with PVL < 200 copies/ml at least during 6 months
* Written informed consent .

Exclusion Criteria:

* Patients with failure to HAART
* Patients with B or C symptoms (CDC classification 1993).
* Age < 18 years old.
* Pregnant or breastfeeding women
* Patients with baseline creatinin > 2.5 mg/dl
* Patients with baseline GOT/GPT > 250 UI/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of steady state viremia (so-called viral set point) after 6-12 months after vaccination with viremia before HAART. | 6 and 12 months

SECONDARY OUTCOMES:
Proportion with evidence of HIV-specific CTL comparing end of immune-based therapy, and end of trial (week 48) with start of immune-based therapy. | 6 and 12 months
Proportion with evidence of HIV-specific T-cell proliferative response comparing end of immune-based therapy, and end of trial (week 48) with start of immune-based therapy. | 6 and 12 months
Proportion with evidence of HIV-specific neutralizing activity of serum comparing end of immune-based therapy, and end of trial (week 48) with start of immune-based therapy. | 6 and 12 months
HIV-1 specific CTL responses in lymphoid tissue | 0 and 6 months
DC Migration | 0 and 2 weeks
Viral load in semen and vaginal secretions | 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Felipe García, MD, PhD, Principal Investigator — Hospital Clínic
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Garcia F, Lejeune M, Climent N, Gil C, Alcami J, Morente V, Alos L, Ruiz A, Setoain J, Fumero E, Castro P, Lopez A, Cruceta A, Piera C, Florence E, Pereira A, Libois A, Gonzalez N, Guila M, Caballero M, Lomena F, Joseph J, Miro JM, Pumarola T, Plana M, Gatell JM, Gallart T. Therapeutic immunization with dendritic cells loaded with heat-inactivated autologous HIV-1 in patients with chronic HIV-1 infection. J Infect Dis. 2005 May 15;191(10):1680-5. doi: 10.1086/429340. Epub 2005 Apr 11. PMID 15838795
- [Result] Garcia F, Climent N, Guardo AC, Gil C, Leon A, Autran B, Lifson JD, Martinez-Picado J, Dalmau J, Clotet B, Gatell JM, Plana M, Gallart T; DCV2/MANON07-ORVACS Study Group. A dendritic cell-based vaccine elicits T cell responses associated with control of HIV-1 replication. Sci Transl Med. 2013 Jan 2;5(166):166ra2. doi: 10.1126/scitranslmed.3004682. PMID 23283367
- [Result] Garcia F, Climent N, Assoumou L, Gil C, Gonzalez N, Alcami J, Leon A, Romeu J, Dalmau J, Martinez-Picado J, Lifson J, Autran B, Costagliola D, Clotet B, Gatell JM, Plana M, Gallart T; DCV2/MANON07- AIDS Vaccine Research Objective Study Group. A therapeutic dendritic cell-based vaccine for HIV-1 infection. J Infect Dis. 2011 Feb 15;203(4):473-8. doi: 10.1093/infdis/jiq077. Epub 2011 Jan 13. PMID 21233310
- [Derived] Andres C, Plana M, Guardo AC, Alvarez-Fernandez C, Climent N, Gallart T, Leon A, Clotet B, Autran B, Chomont N, Gatell JM, Sanchez-Palomino S, Garcia F. HIV-1 Reservoir Dynamics after Vaccination and Antiretroviral Therapy Interruption Are Associated with Dendritic Cell Vaccine-Induced T Cell Responses. J Virol. 2015 Sep;89(18):9189-99. doi: 10.1128/JVI.01062-15. Epub 2015 Jun 24. PMID 26109727
- [Derived] Gil C, Climent N, Garcia F, Hurtado C, Nieto-Marquez S, Leon A, Garcia MT, Rovira C, Miralles L, Dalmau J, Pumarola T, Almela M, Martinez-Picado J, Lifson JD, Zamora L, Miro JM, Brander C, Clotet B, Gallart T, Gatell JM. Ex vivo production of autologous whole inactivated HIV-1 for clinical use in therapeutic vaccines. Vaccine. 2011 Aug 5;29(34):5711-24. doi: 10.1016/j.vaccine.2011.05.096. Epub 2011 Jun 14. PMID 21679735